CLINICAL TRIAL: NCT01735292
Title: Safety of the Automatic Respiration Transfer System- Timer
Acronym: Timer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hadassah Medical Organization (Other)
Collaborators: Shaare Zedek Medical Center (Other)
Responsible Party: Principal Investigator, SPRUNG CHARLES, Director, General Intensive Care Unit, Hadassah Medical Organization
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 0209-12-HMO
Record Dates: First submitted 2012-11-19; First posted 2012-11-28 (Estimated); Last update posted 2012-11-28 (Estimated); Status verified 2012-11

CONDITIONS: Intensive Care Patients on a Ventilator
Keywords: Ventilation, timer
MeSH Terms: conditions — Respiratory Aspiration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Automatic Respiration Transfer System- Timer

SUMMARY:
The Israel Terminally Ill Law, 2005 allows patients who are terminally ill and ventilated to have their ventilator placed on a timer which at a specific time in the future stops the ventilator, maintains the patient on positive pressure (CPAP) and allows the patient not to be reconnected to the ventilator. We will evaluate the safety of the Automatic Respiration Transfer-Timer by assessing vital signs, oxygenation and ventilatory pressures and volumes during the use of the timer with the regular ventilator. In addition, we will evaluate whether the timer stops the ventilator and switches to CPAP at the designated time.

ELIGIBILITY:
Inclusion Criteria:

* Ventilated patients with informed consent

Exclusion Criteria:

* Non- ventilated patients

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2013-01; Primary Completion 2014-01 (Estimated); Study Completion 2014-01 (Estimated)

PRIMARY OUTCOMES:
Safety of the Automatic Respiration Transfer System- Timer | one year
  Number of Adverse Events

CONTACTS AND LOCATIONS:
Overall Officials: Charles Sprung, MD, Principal Investigator — Hadassah Medical Organization
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel, Israel